CLINICAL TRIAL: NCT02799810
Title: Standardized Evaluation of Psychosocial Functioning in Patients Awaiting Lung Transplantation
Brief Title: Psychosocial Evaluation Prior to Lung Transplantation
Acronym: EVALUT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: DZL BREATH-EVALUT
Record Dates: First submitted 2016-04-28; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Lung Transplantation; Psychosomatic Medicine
Keywords: lung transplantation; psychosocial functioning; longitudinal; TERS; adherence; Quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
In a prospective longitudinal cohort study we aim at investigating the extent to which pre-transplant psychosocial levels of functioning predict the medical and psychosocial outcomes of lung transplantation. There is evidence that e.g. persistently elevated depressive symptoms are associated with reduced survival after lung transplantation

DETAILED DESCRIPTION:
There is ample evidence that there are high rates of anxiety and depression among patients with end-stage lung disease. In addition, psychological dysfunction and distress seem to be especially prevalent in patients awaiting lung transplantation. Even though patients benefit from the transplant procedure with respect to long-term health-related quality of life (HRQoL), they also face significant challenges in terms of psychosocial adjustment after the transplantation. There is evidence that e.g. persistently elevated depressive symptoms are associated with reduced survival after lung transplantation.

Currently, the screening process to help select among candidates for organ transplant typically involves considering a variety of psychosocial factors. However, it remains somewhat unclear which criteria are considered important in these evaluations, how differences in various aspects of psychosocial functioning are weighed in making the ultimate decision on the suitability of a patient for transplantation, and the extent to which pretransplant psychosocial characteristics predict the medical and psychosocial outcomes of the procedure. Standardized psychometric instruments with proven reliability and validity can prevent the danger of personal bias in the selection of candidates for transplantation. In addition, structured psychometric instruments can help to identify patients with multiple care needs and can support the development of psychosocial interventions designed to increase quality of life and to decrease the risk of a less favorable transplant outcome through modifying the factors that might place patients at risk.

In a longitudinal prospective cohort study, psychosocial functioning will be assessed at multiple time points both before and after lung transplantation. Assessment of psychosocial functioning will be conducted using a validated, structured interview which allows a comprehensive evaluation of the level of adjustment in 10 aspects of psychosocial functioning - the Transplant Evaluation Rating Scale (TERS) - and standardized self-report instruments. The TERS has shown to be an important and significant predictor of several facets of somatic and psychosocial outcomes e.g. in patients after liver transplantation, left ventricular assist device implantation, and hematopoietic stem cell transplantation.

For each patient, a face-to-face psychosomatic evaluation 1 year after Transplantation will take place during a routine clinical assessments at the Department of Respiratory Medicine.

The following outcome parameters will be assessed:

* Mental disorders (current)
* Psychological processing of lung transplantation (including organ integration and the patient's relationship with the donor, chronic stress/psychological distress and the emotional effects of transplantation/immunosuppression
* Return to work one year after lung transplantation
* Psychological interventions during the first postoperative year
* Intake of (new) psychotropic medication during the first postoperative year

ELIGIBILITY:
Inclusion Criteria:

* patients listed for lung Transplantation (including combined Transplantation) or who are evaluated at the interdisciplinary lung transplant outpatient clinic
* regular post-transplant visits at the Department of Respiratory Medicine
* informed consent

Exclusion Criteria:

* Age below 18 years
* lacking German language skills
* severe cognitive disability
* re-do Transplantation
* colonization with pan- or multi-resistant organisms with Need for isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting for evaluation at the interdisciplinary lung transplant outpatient clinic of Hannover Medical School or already listed for lung Transplantation and being in Treatment at Hannover Medical School
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change in survival status after lung transplantation | assessments at 1, 3, 6 and 12 month after lung transplantation
  number of days survived during first post-operative year

SECONDARY OUTCOMES:
duration of hospitalization after lung transplantation | assessments at 1, 3, 6 and 12 month after lung transplantation
  number of days of hospitalization during first post-operative year
change in adherence during the first post-operative year | assessments at 1, 3, 6 and 12 month after lung transplantation
  mean composite adherence score to immunosuppressants (IS) based on multiple clinical ratings and IS trough levels during first post-operative year
change from baseline quality of life to one year post-transplantation | once before admission to waiting list and 12 month after lung transplantation
  Change in self-rated multidimensional quality of life
change in quality of life during first post-operative year | 1, 3, 6 and 12 month after lung transplantation
  mean self-rated multidimensional quality of life based on multiple assessments during first post-operative year
change from baseline psychological distress (questionnaire) to one year post-transplantation | once before admission to waiting list and 12 month after lung transplantation
  change in levels of self-rated anxiety and depressive symptoms
change in psychological distress (questionnaire) during first post-operative year | 1, 3, 6 and 12 month after lung transplantation
  mean levels of self-rated anxiety and depressive symptoms based on multiple assessments during first post-operative year
mental disorders | 12 month after lung transplantation
  number and kind of current mental disorders at one year after lung transplantation
integration of transplant in own Body Image (questionnaire) | 12 month after lung transplantation
  Quality of psychological processing of lung Transplantation and Feelings towards donor one year after lung transplantation
psychological interventions | 12 month after lung transplantation
  number and kind of psychosocial interventions during first post-operative year
psychotropic medication | 12 month after lung transplantation
  kind and intake of (new) psychotropic medication during first post-operative year
change from baseline comorbidity to one year post-Transplantation (clinical Rating) | once before admission to waiting list and 12 month after lung transplantation
  change in kind, number and degree of comorbid conditions
Change in comorbidity (clinical Rating) | 1, 3, 6 and 12 month after lung transplantation
  mean number and degree of comorbid conditions during first post-operative year

CONTACTS AND LOCATIONS:
Overall Officials: Martina de Zwaan, Prof. Dr., Principal Investigator — Hannover Medical School; Jens Gottlieb, Prof. Dr., Principal Investigator — Hannover Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Gazdag G, Horvath GG, Makara M, Ungvari GS, Gerlei Z. Predictive value of psychosocial assessment for the mortality of patients waiting for liver transplantation. Psychol Health Med. 2016 Jun;21(4):525-529. doi: 10.1080/13548506.2015.1109670. Epub 2015 Nov 7. PMID 26549304
- [Background] Goetzmann L, Irani S, Moser KS, Schwegler K, Stamm M, Spindler A, Buddeberg C, Schmid C, Boehler A, Klaghofer R. Psychological processing of transplantation in lung recipients: a quantitative study of organ integration and the relationship to the donor. Br J Health Psychol. 2009 Nov;14(Pt 4):667-80. doi: 10.1348/135910708X399447. Epub 2009 Jan 24. PMID 19171083
- [Background] Kugler C, Tegtbur U, Gottlieb J, Bara C, Malehsa D, Dierich M, Simon A, Haverich A. Health-related quality of life in long-term survivors after heart and lung transplantation: a prospective cohort study. Transplantation. 2010 Aug 27;90(4):451-7. doi: 10.1097/TP.0b013e3181e72863. PMID 20562734
- [Background] Lowe B, Wahl I, Rose M, Spitzer C, Glaesmer H, Wingenfeld K, Schneider A, Brahler E. A 4-item measure of depression and anxiety: validation and standardization of the Patient Health Questionnaire-4 (PHQ-4) in the general population. J Affect Disord. 2010 Apr;122(1-2):86-95. doi: 10.1016/j.jad.2009.06.019. Epub 2009 Jul 17. PMID 19616305
- [Background] Napolitano MA, Babyak MA, Palmer S, Tapson V, Davis RD, Blumenthal JA; Investigational Study of Psychological Intervention in Recipients of Lung Transplant (INSPIRE) Investigators. Effects of a telephone-based psychosocial intervention for patients awaiting lung transplantation. Chest. 2002 Oct;122(4):1176-84. doi: 10.1378/chest.122.4.1176. PMID 12377839
- [Background] Smith PJ, Blumenthal JA, Carney RM, Freedland KE, O'Hayer CVF, Trulock EP, Martinu T, Schwartz TA, Hoffman BM, Koch GG, Davis RD, Palmer SM. Neurobehavioral functioning and survival following lung transplantation. Chest. 2014 Mar 1;145(3):604-611. doi: 10.1378/chest.12-2127. PMID 24233282
- [Background] Speckhart D, Solomon SR, Zhang X, Morris LE, Bashey A, Holland HK. The Psychosocial Transplant Evaluation Rating Scale (TERS) prospectively predicts inferior Overall survival outcome for high-risk scoring patients undergoing allogeneic hematopoietic stem cell Transplantation. Blood 2014; 124(21)
- [Background] Twillman RK, Manetto C, Wellisch DK, Wolcott DL. The Transplant Evaluation Rating Scale. A revision of the psychosocial levels system for evaluating organ transplant candidates. Psychosomatics. 1993 Mar-Apr;34(2):144-53. PMID 8456157
- [Background] Yost GL, Bhat G, Ibrahim KN, Karountzos AG, Chandrasekaran M, Mahoney E. Psychosocial Evaluation in Patients Undergoing Left Ventricular Assist Device Implantation Using the Transplant Evaluation Rating Scale. Psychosomatics. 2016 Jan-Feb;57(1):41-6. doi: 10.1016/j.psym.2015.07.013. Epub 2015 Aug 1. PMID 26481959